CLINICAL TRIAL: NCT04425863
Title: Evaluation of Ivermectin, Aspirin, Dexamethasone and Enoxaparin as Treatment of covid19
Brief Title: Ivermectin, Aspirin, Dexamethasone and Enoxaparin as Treatment of Covid 19
Acronym: IDEA
Status: Completed | Type: Observational
Sponsor: Eurnekian Public Hospital (Other)
Responsible Party: Principal Investigator, Hector E Carvallo, Principal investigator, Eurnekian Public Hospital
Other Study IDs: IDEA
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Severe Acute Respiratory Syndrome; Ventilation Pneumonitis
Keywords: COVID 19 IVERMECTIN ASPIRIN DEXAMETASONE ENOXAPARIN
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — Ivermectin; Solutions; Aspirin; Ambulatory Care; Dexamethasone; Injections; Hospitalization; Respiration, Artificial; Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Mild cases: This group includes patients diagnosed positive for COVID-19 via rtPCR and presenting only mild symptoms such as: fever not above 38.5 °C; isolated diarrheal episodes, hyposmia or hypogeusia, mild desaturation (93 - 96 %), dyspnea without matter, polymyoarthralgias, persistent headache, abdominal pain.
  Interventions: Drug: Ivermectin 5 MG/ML oral solution, Aspirin 250 mg tablets
- Moderate cases: This group includes patients diagnosed positive for COVID-19 via rtPCR and presenting either: 3 severe symptoms (i.e. fever above 38.5 °C, diarrhea with more than 3 daily depositions, flictenular conjunctivitis, strong desaturation (92% or less), tachypnea (FR> 25 / minute) or 2 severe symptoms + 2 mild symptoms (fever not above 38.5 °C; isolated diarrheal episodes, hyposmia or hypogeusia, mild desaturation (93 - 96 %), dyspnea without matter, polymyoarthralgias, persistent headache, abdominal pain)
  Interventions: Other: Ivermectin 5 mg/mL oral solution, Dexamethasone 4-mg injection, Aspirin 250 mg tablets
- Severe cases: This group includes patients diagnosed positive for COVID-19 via rtPCR and presenting either: 4 severe symptoms or 3 severe symptoms and not less than 2 mild symptoms or clinical signs of bilateral viral pneumonia
  Interventions: Other: Ivermectin 5 MG/ML oral solution, Dexamethasone 4-mg injection, Enoxaparin injection. Inpatient treatment with mechanical ventilation in ICU.

INTERVENTIONS:
Drug: Ivermectin 5 MG/ML oral solution, Aspirin 250 mg tablets — 24 mg oral Ivermectin on days 0 and 7 and 1 Aspirin tablet daily for 30 days. Outpatient treatment.
  Other Names: Outpatient treatment
  Groups: Mild cases
Other: Ivermectin 5 mg/mL oral solution, Dexamethasone 4-mg injection, Aspirin 250 mg tablets — 36 mg oral Ivermectin on days 0 and 7; 1 daily injection of 4-mg Dexamethasone until discharge, 1 Aspirin tablet daily for 30 days. Inpatient treatment in ward care, including Low flow washed oxygen or oxygen concentrator
  Other Names: Inpatient treatment in ward care
  Groups: Moderate cases
Other: Ivermectin 5 MG/ML oral solution, Dexamethasone 4-mg injection, Enoxaparin injection. Inpatient treatment with mechanical ventilation in ICU. — 48 mg oral Ivermectin on days 0 and 7; 1 daily injection of 4-mg Dexamethasone until discharge, Enoxaparin 100 IU/kg (ca. 1 mg/kg) daily until transfer to ward care. Then continue with inpatient treatment in ward care.
  Other Names: Inpatient treatment in ICU
  Groups: Severe cases

SUMMARY:
The associated use of Ivermectin, aspirin, dexamethasone, and enoxaparin (in different combinations and doses) will reduce the impact of COVID infection 19, the need of admission to the intensive care unit, and mortality.

DETAILED DESCRIPTION:
Between 30 and 50% of patients who contract COVID 19 will be asymptomatic or oligosymptomatic. This fact will not give rise to the consult, and will directly affect a notorious sub-registration of the cases.

The second, even more disturbing, premise is that these patients are as contagious as the moderate and severe cases.

The virus incubation period has been calculated at 5.1 days (95% CI, 4.5 to 5.8 days), and 97.5% of patients are said to have symptoms at 11 days (95% CI 8.2 to 15.6 days).

A mortality of 5.7% has been calculated. The average COVID patient presents with fever (78%), cough (60-79%) and myalgias or fatigue (35.8 to 44%).

55% develop dyspnea, which appears on average 8 days after the onset of symptoms.

To the manifestations expressed above, the presence of bilateral conjunctival injection should be added, without associated secretions, hypogeusia, skin rash and hyposmia.

Diagnostic confirmation is made through laboratory studies, which can be performed on a wide variety of biological samples.

Bronchoalveolar lavage samples showed the highest sensitivity (93%), followed by sputum samples (72%), nasal swabs (63%), fiberoptic brush biopsy (46%), pharyngeal swabs (32%), feces ( 29%) and, finally, blood (1%). A sensitivity of 91% is reported in saliva samples.

Evidence suggests that a subgroup of patients with severe forms of COVID 19 may have cytokine storm syndrome.

Therefore, we recommend the identification and treatment of hyperinflammation using existing approved therapies with proven safety profiles to address the immediate need to reduce increasing mortality (see Therapeutic Proposal).

Secondary hemophagocytic lymphohistiocytosis (SHLH) is a poorly recognized hyperinflammatory syndrome characterized by fatal and fulminant hypercytokinemia with multiple organ failure.

In adults, SHLH is most often triggered by viral infections, and occurs in 3.7-4.3% of sepsis cases.

The cardinal features of sHLH include constant fever, cytopenias, and hyperferritinemia; Pulmonary involvement (including ARDS) occurs in approximately 50% of patients.

A cytokine profile that resembles sHLH is associated with the severity of COVID-19 disease, characterized by an increase in interleukin (IL) -2, IL-7, granulocyte colony stimulating factor, protein 10 inducible by interferon-γ, monocyte chemoattractant protein, macrophage inflammatory protein 1-α and tumor necrosis factor-α.

Mortality predictors from a recent multicenter retrospective study of 150 confirmed cases of COVID-19 in Wuhan, China included elevated ferritin (mean 1297.6 ng / ml in non-survivors versus 614.0 ng / ml in survivors; p <0.001) and IL-6 (p <0.0001), suggesting that mortality could be due to viral hyperinflammation.

However, cases have been reported where tissue and organ involvement has been found whose concentration of ACE receptors is very dissimilar (myocardium, brain). In all of them, the common denominator was small vessel thrombosis, as seen in entities such as Catastrophic Antiphospholidic Syndrome.

Currently the Virchow triad factors have been narrowed down in more detail:

Circulatory stasis: abnormalities of hemorrheology and turbulence in vascular bifurcations and stenotic regions.

Injury to the vascular wall: abnormalities in the endothelium, such as atherosclerosis and associated vascular inflammation.

Hypercoagulable state: abnormalities in the coagulation and fibrinolytic pathways and in platelet function associated with an increased risk of VTE and other cardiovascular diseases (such as coronary artery disease [CPA], heart failure and stroke in patients with AF). All lead to a state of hypercoagulability, which could explain the formation of microthrombosis in different locations, as has been repeatedly reported in patients with COVID 19.

BASES OF THE PROPOSED THERAPEUTICS They rest on four pillars: Ivermectin, Aspirin, Dexamentasone and Enoxaparin. IVERMECTIN Ivermectin is a broad-spectrum antiparasitic, with vermicidal and ectoparasiticidal properties. It was discovered and marketed for animal use in the early 1980s.

Approved in 1997 by the FDA for single-dose strongyllidiasis of 200 mcg / kg and crusted scabies (Scabies Norway) in patients with AIDS at a dose of 200 mcg / kg, every week for 2 weeks.

In Argentina, it has been available for human use for almost 20 years. But, much more recently, its viricidal effects have been compiled on different varieties of flavivirus, dengue, Zica, Chikunguña, etc.

Ivermectin has been reported to be a SARS-CoV-2 inhibitor. This activity is believed to be due to the dependence of many different RNA viruses on IMPα / β1 during infection. These reports suggested that the inhibitory activity of ivermectin nuclear transport may be effective against SARS-CoV-2, since they demonstrate that ivermectin has antiviral action against the clinical isolate of SARS-CoV-2 in vitro, with a single dose capable to control viral replication in 24-48 hours. in vitro.

Although in vitro studies have used doses that -extrapolated to those recommended in the treatment of ectoparasitosis in humans- might seem high, the truth is that studies carried out in healthy volunteers, more than two decades ago, proved that the usual doses they can be increased tenfold, without significant side and / or adverse effects.

ASPIRIN Aspirin is the common name for acetylsalicylic acid. The chemical production is based on the salicylic acid obtained by synthesis. Its most common uses and for what it was first used was as an analgesic (for pain), antipyretic (to lower fever) and anti-inflammatory. It is classified as a non-steroidal anti-inflammatory drug (NSAID). In 1989 the first large study was published that proved that Aspirin reduces cardiovascular risk, acting as an antiplatelet agent.

These were low-dose Aspirin, and the risk of myocardial infarction was found to decrease by 44% when the previously named dose of Aspirin was administered.

HEPARIN AND ENOXAPARIN Heparins are injectable anticoagulant substances. A distinction should be made between standard heparin or unfractionated heparin (HNF) and low molecular weight heparins (LMWH).

HNF is made up of a heterogeneous mixture of polysaccharide chains of variable length.

LMWHs are the result of fragmentation of HNF by different methods to achieve products with lower and more homogeneous molecular weights. They are also made up of a mixture of polysaccharide chains and their average molecular weight is much lower. The antithrombotic and anticoagulant activity of HNF is related to the ability to inhibit factor Xa and factor IIa respectively. LMWHs have less inhibitory activity to thrombin or factor IIa but maintain the same potency with respect to factor Xa, so it is expected that they present a lower risk of bleeding but the same antithrombotic activity.

CORTICOSTEROIDS Systemic corticosteroids are powerful anti-inflammatory and immunosuppressive agents. They can be administered intravenously, intramuscularly, orally, intralesionally, and topically. Its side effects increase with high, long and frequent doses. Corticosteroids are drugs frequently used in various clinical situations, because they are powerful anti-inflammatories and immunomodulators. Glucocorticoids passively diffuse through the cell membrane, then join soluble receptor proteins in the cytoplasm. They are used, among others, for the treatment of some rheumatic diseases. A separate case, well known but not studied in the current contingency, is acute adrenal insufficiency.

CURRENT IDEA TRIAL Based on the precedent data, we started a Clinical Trial based on the above-mentioned four drugs, on a gradual scale, and according the severity of each case. In order to determine the dose and combination, we developed our own Severity Score.

INTERPRETATION:

Mild cases Only minor criteria findings Moderate cases 3 major crit. findings, or 2 major + 2 minor Severe cases 4 major crit. Findings or 3 major + 2/3 minor

Based on the previous criteria, we used the following combinations and doses:

DISEASE SEVERITY Firm Suspicious Case or Confirmed case 24 mg orally at a dose of 200 ug / kg in a single dose, to be repeated a week later Aspirin 250 mg orally Moderate clinical stage 36 mg orally at a dose of 400 ug / kg in a single dose, to be repeated a week later Dexamethasone 4 mg/day (parenteral) Aspirin 250 mg orally Low Flow Washed Oxygen or Oxygen Concentrator Severe case with bilateral pneumonia 48 mg via gastric cannulae, to be repeated a week later Dexamethasone 4 mg/day (parenteral) Enoxaparin100 UI/kg (1 mg/kg) Mechanical Ventilation

ELIGIBILITY:
Inclusion Criteria:

patients with positive oral/nasal swabs

Exclusion Criteria:

Children under 5 years old Pregnant women Previous reports of allergy to any of the drugs used in the clinical trial

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients bothe genders, ages 5 or up, non pregnant, capable of accepting participation in trial (granted by signed premission), and affected by COVID 19
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Secchi, M.D., Study Chair — President Ethical Commitee, Hospital Eurnekian
Locations (1):
- Hospital Eurnekian, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
Personal data will remain secret. Only clinical descriptions (age, gender, co-morbidities, evolution, outcomes will be released

REFERENCES:
- [Background] Rizzo E. Ivermectin, antiviral properties and COVID-19: a possible new mechanism of action. Naunyn Schmiedebergs Arch Pharmacol. 2020 Jul;393(7):1153-1156. doi: 10.1007/s00210-020-01902-5. Epub 2020 May 27. PMID 32462282
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at Eurnekian Public Hospital
Groups:
- Moderate Cases: This group includes patients diagnosed positive for COVID-19 via rtPCR an presenting either: 3 severe symptoms (i.e. fever above 38.5 °C, diarrhea with more than 3 daily depositions, flictenular conjuntivitis, strong desaturation of 92 % or less, tachypnea with FR higher than 25/minute) or 2 severe symptoms + 2 mild symptoms (as already described for mild cases).
Period: Overall Study
Arm/Group | Mild Cases | Moderate Cases | Severe Cases
Started | 135 | 12 | 20
Completed | 135 | 12 | 19
Not Completed | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Mild Cases: Patients diagnosed positive for COVID-19 and presenting only mild symptoms.
- Moderate Cases: Patients diagnosed positive for COVID-19 and presenting either 3 severe symptoms or 2 severe symptoms + 2 mild symptoms
- Severe Cases: Patients diagnosed positive for COVID-19 and presenting either 4 severe symptoms or 3 severe symptoms + not less than 2 mild symptoms or clinical symptoms of bilateral viral pneumonia
- Total: Total of all reporting groups
Arm/Group | Mild Cases | Moderate Cases | Severe Cases | Total
Number analyzed (Participants) | 135 | 12 | 20 | 167
Age, Continuous [Mean (Full Range); unit: years] | 55.7 [41 to 88] | 59.7 [41 to 88] | 59.7 [41 to 88] | 56.5 [41 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 7 | 11 | 84
  Male | 69 | 5 | 9 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 135 | 12 | 20 | 167
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 135 | 12 | 20 | 167
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 135 | 12 | 20 | 167

OUTCOME MEASURES:

1. Primary Outcome: Patients Who Improved Their Condition or Did Not Worsen it
Description: Number of patients who did not go to a more severe stage of disease or die (i.e. they neither go from mild to moderate or severe, nor go from moderate to severe or die, if they had been already enrolled in a severe condition)
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Mild Cases: Patients diagnosed positive for COVID-19 via rtPCR and presenting only mild symptoms. No clinical signs of viral pneumonia.
- Moderate Cases: Patients diagnosed positive for COVID-19 and presenting either 3 severe symptoms or 2 severe symptoms + 2 mild symptoms. Clinical sign of viral pneumonia.
- Severe Cases: Patient diagnosed positive for COVID-19 presenting 4 severe symptoms or 3 severe symptoms and not less than 2 mild symptoms. Clinical signs of bilateral viral pneumonia.
Arm/Group | Mild Cases | Moderate Cases | Severe Cases
Number analyzed (Participants) | 135 | 12 | 20
Participants | 135 | 12 | 19

2. Primary Outcome: ICU-treated Patients After 2-week Treatment
Description: Number of patients needing ICU-treatment including mechanical ventilation after 2-week treatment
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Groups:
- Mild Cases: Patients diagnosed positive for COVID-19 via rtPCR, presenting only mild symptoms and no clinical sign of viral pneumonia.
- Moderate Cases: Patients diagnosed positive for COVID-19 via rtPCR, presenting either 3 severe symptoms or 2 mild severe symptoms + 2 mild symptoms or clinical signs of viral pneumonia.
- Severe Cases: Patients diagnosed positive for COVID-19, presenting either 4 severe symptoms or 3 severe symptoms + at least 2 mild symptoms or clinical signs of bilateral viral pneumonia
Arm/Group | Mild Cases | Moderate Cases | Severe Cases
Number analyzed (Participants) | 135 | 12 | 20
Participants | 0 | 0 | 2

3. Primary Outcome: Mortality
Description: Patients who died within 30 days after enrollment
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Mild Cases: Patients diagnosed positive for COVID-19 presenting only mild symptoms and no clinical signs of viral pneumonia.
- Moderate Cases: Patients diagnosed positive for COVID-19 and presenting either 3 severe symptoms or 2 severe + 2 mild symptoms and showing clinical signs of viral pneumonia.
- Severe Cases: Patients diagnosed positive for COVID-19 and presenting either 4 severe symptoms or 3 severe symptoms + 2 mild symptoms or clinical signs of bilateral viral pneumonia.
Arm/Group | Mild Cases | Moderate Cases | Severe Cases
Number analyzed (Participants) | 135 | 12 | 20
Participants | 0 | 0 | 1
Statistical Analysis 1: Comparison: Moderate Cases vs Severe Cases; A chi-squared test is used to find out whether there is a statistically significant decrease in mortality rate when the IDEA treatment protocol is used in hospitalized patients in comparison with other treatments in the same hospital in the same period of time (3 out of 12 inpatients died); Test type: Other; p = 0.0246, Chi-squared
Statistical Analysis 2: Comparison: Mild Cases vs Moderate Cases vs Severe Cases; Overall mortality rate of patients treated according to IDEA protocol is compared by a chi-squared test against overall mortality rate in Argentina (the same region where the hospital is located). Data used for overall mortality in Argentina correspond to June 30th according to the website of the Ministry of Health of Argentina; Test type: Other; p = 0.0475, Chi-squared
Statistical Analysis 3: Comparison: Moderate Cases vs Severe Cases; A chi-square test was applied to compare the mortality rate of patients treated with IDEA protocol as compared with data published (26.84 %) in Bertsimas D, Lukin G, Mingardi L, Nohadani O, Orfanoudaki A, Stellato B et al. (2020), COVID-19 Mortality Risk Assessment: An International Multi-Center Study doi: 10.1101/2020.07.07.20148304; Test type: Other; p = 0.0025, Chi-squared

4. Primary Outcome: Patients Needing Drug Dose Adjustment
Description: Patients who needed dose adjustment of any of the drugs involved in the treatment protocol
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Groups:
- Mild Cases: Patients diagnosed positive for COVID-19 presenting only mild symptoms and no clinical sign of viral pneumonia.
- Moderate Cases: Patients diagnosed positive for COVID-19 by rtPCR and presenting 3 severe symptoms or 2 mild + 2 severe symptoms or clinical signs of viral pneumonia.
- Severe Cases: Patients diagnosed positive for COVID-19 by rtPCR and presenting 4 severe symptoms or 3 severe symptoms + 2 mild symptoms or clinical signs of bilateral viral pneumonia.
Arm/Group | Mild Cases | Moderate Cases | Severe Cases
Number analyzed (Participants) | 135 | 12 | 20
Participants | 0 | 0 | 0

5. Primary Outcome: Adverse Events
Description: Patient presenting serious adverse events
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Groups:
- Mild Cases: Patients diagnosed positive for COVID-19 by rtPCR and presenting only mild symptoms and no clinical sign of viral pneumonia.
- Moderate Cases: Patients diagnosed positive for COVID-19 by rtPCR and presenting either 3 severe symptoms or 2 severe symptoms + 2 mild symptoms or clinical signs of viral pneumonia.
- Severe Cases: Patients diagnosed positive for COVID-19 by rtPCR, presenting 4 sever symptoms, or 3 severe symptoms + 2 mild symptoms or clinical signs of bilateral viral pneumonia.
Arm/Group | Mild Cases | Moderate Cases | Severe Cases
Number analyzed (Participants) | 135 | 12 | 20
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Moderate Cases: Patients diagnosed positive for COVID-19 by rtPCR presenting 3 severe symptoms or 2 severe symptoms + 2 mild symptoms or clinical signs of viral pneumonia
- Severe Cases: Patients diagnosed positive for COVID-19 by rtPCR presenting 4 severe symptoms or 3 severe symptoms + 2 mild symptoms or clinical signs of bilateral viral pneumonia
Arm/Group | Mild Cases | Moderate Cases | Severe Cases
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/12 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/12 | 1/20
Other Adverse Events (participants affected / at risk) | 0/135 | 0/12 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Cases (N=135) | Moderate Cases (N=12) | Severe Cases (N=20)
multiple organ failure (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Multiple organ failure and respiratory defficiency leading to death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Cases (N=135) | Moderate Cases (N=12) | Severe Cases (N=20)
Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Required only minor intervention. The patient had an ulcer at enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT04425863/Prot_SAP_000.pdf